CLINICAL TRIAL: NCT04614207
Title: Predictors of Physical Activity Levels in Children and Adolescents With Cerebral Palsy - a Clinical Cohort Study
Brief Title: Cerebral Palsy & Predictors of Physical Activity
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Elsass Foundation (Other); Region of Southern Denmark (Other); AJ Andersen og Hustrus Fond (Other); The Hede Nielsen Family Foundation (Other); Dagmar Marshalls Fond (Unknown); Fonden til Lægevidenskabens Fremme (Other)
Responsible Party: Sponsor
Other Study IDs: 1-Fonvig
Record Dates: First submitted 2020-11-02; First posted 2020-11-03 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Cerebral Palsy
Keywords: Physical activity; Accelerometry; Quality of life; Children; Adolescents
MeSH Terms: conditions — Cerebral Palsy; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Children and adolescents with cerebral palsy may be trapped in a vicious circle of low physical fitness, early fatigue in daily activities, resulting in deconditioning and a further decrease in physical activity. From this perspective, establishing a healthy and active lifestyle during childhood is even more important for individuals with a disability, who are at higher risk for functional limitations and general fatigue in addition with developing secondary' conditions such as cardiovascular disease, diabetes, and obesity. Furthermore, physical activity has a positive impact on quality of life, but it remains unknown which factors that influence high levels of habitual physical activity in children and adolescents with cerebral palsy.

The present research project will investigate predictors of habitual physical activity in children and adolescents with cerebral palsy with the perspective of providing evidence on optimizing physical activity and consequently improved overall health.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a condition that describes a group of disorders (altered muscle tone, movements disorder, muscle weakness, ataxia and rigidity) covering the development of movement and posture causing activity limitations and reduced quality of life (1). In Denmark 2000-2500 children and adolescents under the age of 18 are living with the diagnosis of cerebral palsy. This is equivalent to two children being diagnosed with cerebral palsy per 1000 living births (2). Though, CP is a non-progressive diagnosis, it is a lifelong condition that requires attention through most of the patient's life, as impairments that inhibit performance of activities and participation in daily living develops (1, 3). Children and adolescents with cerebral palsy are a vulnerable group who find it challenging to meet the physical activity guidelines, therefore predisposing them to the negative health implications associated with low levels of physical activity and high levels of sedentary time (4).

Although there are no specific evidence-based physical activity guidelines for children and adolescents with cerebral palsy, it is clear that they have lower levels of physical activity than their peers, that they do not meet the World Health Organization's physical activity guidelines, and that their level of mobility limitation is negatively associated with their level of physical activity (5, 6).

Therefore, the objective of this study is to investigate predictors of physical activity and inactivity in children and adolescents with cerebral palsy with the perspective of providing evidence-based motivators for optimized physical activity, with the potential benefit of improved overall health and quality of life.

This is a prospective clinical cohort study. Eligible children and adolescents and their families will be identified through the Danish Health Data Authority after which the parents/guardians will receive written information about the study through digital post, e-Boks.

Parents/guardians will be asked to fill out questionnaires on quality of life, overall health, pain and participation in normal daily activities, and the children/adolescents will be asked to wear accelerometers for seven consecutive days. Data from the Cerebral Palsy FollowUp Program (CPUP) register will be collected.

The project will be implemented in accordance with the Helsinki Declaration II. It has been approved by the Danish Data protection Agency and has been declared not notifiable by the Regional Committee on Health Research Ethics, cf. Committee Act Art. 14, paragraph 1 (S-20192000-23). All subject data will be treated confidentially and in confidence under the Danish laws on personal data and health.

This study will provide novel evidence that will improve the knowledge on how to optimize physical activity, and thus improve overall health and quality of life, for the current group of children and adolescents. Due to wide inclusion criteria, this knowledge will constitute a high level of generalizability and most probably high acceptance by the treating health professionals as the majority of variables of interest already are implemented in a current cerebral palsy registry. Finally, the findings may be implemented in evidence-based physical activity guidelines, which currently are lacking for the present group of children and adolescents with cerebral palsy.

1. Koman LA, Smith BP, Shilt JS. Cerebral palsy. Lancet (London, England). 2004;363(9421):1619-31.
2. Frøslev-Friis C, Dunkhase-Heinl U, Andersen JD, Stausbøl-Grøn B, Hansen AV, Garne E. Epidemiology of cerebral palsy in Southern Denmark. Danish medical journal. 2015;62(1):A4990.
3. Bell KJ, Ounpuu S, DeLuca PA, Romness MJ. Natural progression of gait in children with cerebral palsy. J Pediatr Orthop. 2002;22(5):677-82.
4. Organization WHO. Global recommendations for physical activity for health. Switzerland2010.
5. Carlon SL, Taylor NF, Dodd KJ, Shields N. Differences in habitual physical activity levels of young people with cerebral palsy and their typically developing peers: a systematic review. Disability and rehabilitation. 2013;35(8):647-55.
6. Bjornson KF, Belza B, Kartin D, Logsdon R, McLaughlin JF. Ambulatory physical activity performance in youth with cerebral palsy and youth who are developing typically. Phys Ther. 2007;87(3):248-57.

ELIGIBILITY:
Inclusion Criteria:

* Children born in the timeperiod 2003 - 2013
* Diagnosed with cerebral palsy (according to current classifications)
* Gross Motor Function Classification System (GMFCS) level I - III
* Registered in the Cerebral Palsy Follow-up Registry (CPUP), Denmark (As explained in the Statistical Analysis Plan dated June 6, 2022, CPUP data will be used were available. However, being registred in the CPUP database is no longer a requirement).

Exclusion criteria:

- Parents/guardians unable to read and understand Danish.

Ages: 8 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: All children and adolescents between the ages of 8 and 15 years, diagnosed with cerebral palsy in Denmark. The study population will be selected thru the Danish Health Data Authority ('Sundhedsdatastyrelsen') where social security numbers of parents/guardians sharing an adresse with an individual from the study population, will be used as a means of contact.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Model 1a: Prediction of habitual physical activity using data from the CPUP registry | Response variable is measured between 0 and 39 months post registry data (predictive variables).
  Habitual physical activity will be assessed objectively using accelerometer counts.
  Multiple linear regression analyzes between accelerometer counts (response variable) and all CPUP variables within each ICF (International Classification of Functioning, Disability and Health) component as predictive variables, using the latest CPUP registration prior to accelerometer data collection.

SECONDARY OUTCOMES:
Model 1b: Prediction of habitual physical activity using data from questionnaire variables | Response variable is measured between 1 and 15 months post registry data (predictive variables).
  Habitual physical activity will be assessed objectively using accelerometer counts.
  Multiple linear regression analysis between accelerometer counts (response variable) and all questionnaire variables within each ICF component (predictive variables), using the questionnaire data.
Model 2a: Prediction of habitual physical activity using data from the CPUP registry (penalized regression) | Response variable is measured between 0 and 39 months post registry data (predictive variables).
  Penalized regression (lasso) with accelerometer counts as the response variable and covariates as chosen by lasso to obtain an optimal fit from model 1a as predictive variables to determine which variables to retain in the model.
Model 2b: Prediction of habitual physical activity using data from questionnaire variables (penalized regression) | Accelerometer data is collected 1-15 months post collection of questionnaire data.
  Penalized regression (lasso) with accelerometer counts as the response variable and covariates as chosen by lasso to obtain an optimal fit from model 1b as predictive variables to determine which variables to retain in the model.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Holsgaard-Larsen, Assoc. Prof, Study Director — Department of Clinical Research, University of Southern Denmark.; Christina E Fonvig, MSc, Principal Investigator — Department of Clinical Research, University of Southern Denmark.
Locations (1):
- University of Southern Denmark, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to ethical and legal considerations, our data cannot be shared publicly. This is due to the restrictions from the Regional and the National Committee on Health Research Ethics and the General Data Protection Regulation (EU) 2016/679, since the data contains person-specific information on sex, birth date, and cerebral palsy classification among other.
  Data are available for researchers who meet the criteria for access to confidential data. Access may be acquired through contact to the research group.

REFERENCES:
- [Derived] Fonvig CE, Troelsen J, Dunkhase-Heinl U, Lauritsen JM, Holsgaard-Larsen A. Predictors of physical activity levels in children and adolescents with cerebral palsy: clinical cohort study protocol. BMJ Open. 2021 Sep 21;11(9):e047522. doi: 10.1136/bmjopen-2020-047522. PMID 34548350

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/07/NCT04614207/Prot_SAP_001.pdf